CLINICAL TRIAL: NCT02006381
Title: Ontogenic Measurement of Plasma Oxytocin in Typically Developing Boys Using Extracted and Unextracted EIA Methods
Brief Title: Oxytocin Levels in Typically Developing Boys
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Linmarie Sikich, MD, Associate Professor of Psychiatry, University of North Carolina, Chapel Hill
Other Study IDs: 13-3288
Record Dates: First submitted 2013-11-22; First posted 2013-12-10 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Boys
Keywords: healthy boys; plasma oxytocin; pediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Age 3-6: This will include 10 typically developing boys age 3-6
- Age 7-12: This will include 10 typically developing boys age 7-12
- Age 13-17: This will include 10 typically developing boys age 13-17

SUMMARY:
Measuring basal levels of plasma oxytocin in individuals with typical development across childhood and adolescence using both extracted and unextracted EIA methods.

DETAILED DESCRIPTION:
Measuring basal levels of plasma oxytocin in individuals with typical development across childhood and adolescence using both extracted and unextracted EIA methods. This study is necessary since there is great variability in reported plasma oxytocin in typically developing children from other studies as well as up to 1000 fold variability in such levels using different assay procedures. Further existing studies have not clearly described variation in levels with age. all samples will be taken in the afternoon.

ELIGIBILITY:
Inclusion Criteria:

* Between 3 and 17 years old, inclusive
* Consent of parent or guardian.

Exclusion Criteria:

* Exclusion Criteria for Healthy Control Participants:
* Female gender
* Evidence of a mental health diagnosis
* Evidence of significant medical condition (ie: renal, cardiovascular or genetic disease)
* First degree family member with an ASD diagnosis

Ages: 3 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This population will be a community sample representative of the community of the area.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Plasma Oxytocin Levels | Baseline oxytocin level at visit 1 (time zero)
  20 children in each of 3 age cohorts 3-6, 7-12, and 13-17 will participate. Plasma oxytocin levels will be taken at the screening appointment.

SECONDARY OUTCOMES:
Inflammatory markers | at single time point
  C reactive protein and cytokine panel

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States